CLINICAL TRIAL: NCT03754985
Title: Hyperbaric Oxygen Therapy Effects on Pulmonary Functions
Acronym: PulmHBOT
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0024-16-ASF
Record Dates: First submitted 2018-11-25; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Oxygen Toxicity; Hyperoxia
MeSH Terms: conditions — Hyperoxia | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Hyperbaric Oxygen Therapy: The study included participants 18 years or older, scheduled for 60 HBOT sessions for any indication.
  Interventions: Device: Hyperbaric oxygen therapy

INTERVENTIONS:
Device: Hyperbaric oxygen therapy — The study included participants 18 years or older, scheduled for 60 HBOT sessions for any indication.
  After signing an informed consent form, the participants underwent a pulmonary function baseline evaluation. Participants were treated in a multiplace chamber (HAUX-Life-Support GmbH) for 60 daily sessions, 5 days a week. Each session consisted of 90 minutes of exposure to 100% oxygen at 2 ATA with 5 minute air breaks every 20 minutes. Participants repeated their pulmonary function evaluation after the last HBOT session.
  After signing an informed consent form, the participants underwent a pulmonary function baseline evaluation. Participants were treated in a multiplace chamber (HAUX-Life-Support GmbH) for 60 daily sessions, 5 days a week. Each session consisted of 90 minutes of exposure to 100% oxygen at 2 ATA with 5 minute air breaks every 20 minutes. Participants repeated their pulmonary function evaluation after the last HBOT session.

SUMMARY:
Prospective analysis included patients, 18 years or older, scheduled for 60 daily HBOT sessions between 2016-2018. Each session was 90 min of 100% oxygen at 2 ATA with 5 minutes air breaks every 20 min, five days per week. Pulmonary functions,measured at baseline and after HBOT,included forced vital capacity (FVC), forced expiratory volume in one second (FEV1), peak expiratory flow rate (PEF).

DETAILED DESCRIPTION:
After signing an informed consent form, the participants underwent a pulmonary function baseline evaluation. Participants were treated in a multiplace chamber (HAUX-Life-Support GmbH) for 60 daily sessions, 5 days a week. Each session consisted of 90 minutes of exposure to 100% oxygen at 2 ATA with 5 minute air breaks every 20 minutes. Participants repeated their pulmonary function evaluation after the last HBOT session.

Pulmonary function Measurements of pulmonary functions were performed using the MiniSpir testing apparatus (MIR- Medical International Research, USA). The equipment was calibrated using a 3-liter syringe before performing measurements according to the manufacturer's instructions. Measurements were performed by a trained technician. The forced expiratory maneuvers were performed as recommended by the guidelines[13].

The forced vital capacity (FVC), forced expiratory volume in one second (FEV1) and peak expiratory flow rate (PEF) were taken as the highest readings obtained from at least three satisfactory forced expiratory maneuvers. Mean forced mid-expiratory flow rate (FEF25-75%) and forced expiratory flow rates at 25, 50 and 75% of FVC expired (FEF25%, FEF50% and FEF75%) were taken as the best values from flow-volume loops not differing by >5% from the highest FVC.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older patients
* scheduled for 60 HBOT sessions for any indication

Exclusion Criteria:

* Active smokers were excluded but patients who quit smoking more than six months prior to inclusion were allowed in the study.
* active smoking
* severe known pulmonary disease
* chest pathology incompatible with HBOT
* inner ear disease
* claustrophobia
* other neurological conditions
* pregnancy
* previous HBOT within six months prior to inclusion
* the inability to sign informed consent.

Age Groups: Child, Adult, Older Adult
Study Population: The study included participants 18 years or older, scheduled for 60 HBOT sessions for any indication
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
forced vital capacity (FVC) | change within 3 months
forced expiratory volume in one second (FEV1) | change within 3 months
peak expiratory flow rate (PEF) | change within 3 months
forced mid-expiratory flow rate (FEF25-75%) | change within 3 months
FEV1/FVC ratio | change within 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Amir Hadanny, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Amir Hadanny, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hadanny A, Zubari T, Tamir-Adler L, Bechor Y, Fishlev G, Lang E, Polak N, Bergan J, Friedman M, Efrati S. Hyperbaric oxygen therapy effects on pulmonary functions: a prospective cohort study. BMC Pulm Med. 2019 Aug 13;19(1):148. doi: 10.1186/s12890-019-0893-8. PMID 31409407